CLINICAL TRIAL: NCT00753116
Title: Renal Denervation in End Stage Renal Disease Patients With Refractory Hypertension
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medtronic Vascular (Industry)
Responsible Party: Craig Straley, Ardian Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TP-041
Record Dates: First submitted 2008-09-12; First posted 2008-09-16 (Estimated); Last update posted 2012-11-06 (Estimated); Status verified 2012-11

CONDITIONS: Kidney Failure, Chronic; Renal Dialysis
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Renal Denervation with a catheter-based procedure — Disruption of the renal nerves with a catheter-based procedure

SUMMARY:
The purpose of this this study is to investigate the clinical utility of renal denervation in the treatment of ESRD patients with refractory hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Systolic blood pressure of 160 mmHg or greater
* On 3 or more antihypertensive medications
* On dialysis for more than 6 months

Exclusion Criteria:

* Renal artery abnormalities
* Known secondary hypertension attributable to a cause other than sleep apnea
* MI, angina, CVA within 6 months
* Others

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2008-09; Primary Completion 2008-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Safety - complications associated with delivery and/or use of the Ardian Catheter, adverse renal events, electrolyte disturbances, hemodynamic events. | Through 1 year

SECONDARY OUTCOMES:
Physiologic response to denervation (e.g., blood pressure reduction) | Through 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Hennepin County Medical Center, Minneapolis, Minnesota, United States